CLINICAL TRIAL: NCT03923413
Title: Endothelial Function and Circulating Microparticle in Patients Under LVAD Support
Acronym: MP-LVAD
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Dr.med. Patrick Horn, Principle Investigator, Heinrich-Heine University, Duesseldorf
Other Study IDs: 14-018
Record Dates: First submitted 2019-04-12; First posted 2019-04-22 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: End Stage Heart Failure
Keywords: circulating MP; FMD; LVAD; endothelial function; endothelial integrity
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3ml venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with chronic heart failure without LVAD support: patients with chronic heart failure without LVAD support
  Interventions: Other: Blood samples
- patients with end-stage heart failure with LVAD support: patients with end-stage heart failure with LVAD support
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples for MP evaluation

SUMMARY:
The aims of this project are 1) to evaluate whether circulating micraparticals (MPs) in patients with LVAD impair endothelial function and 2) to assess the procoagulative activity of circulating MPs in patients with LVAD in a prospective longitudinal study of patients undergoing LVAD implantation, 3) to analyze these parameters in the context of thromboembolic events.

DETAILED DESCRIPTION:
Continuous-flow left ventricular assist devices (LVADs) have arised as a vital therapeutic option in end stage heart failure not merely as bridge-to transplant but also as destination therapy. LVADs are associated with impaired endothelial function as well as with a dysbalance of coagulation leading to both, excessive bleeding and thromboembolic events, respectively. Microparticles (MPs) are shed membrane particles budded into the circulation and considered as a marker of compromised endothelial integrity and enhanced procoagulation levels. In addition, MPs have been suggested to play an active role in the induction of endothelial dysfunction and coagulation. First studies demonstrated increased level of MPs in patients with LVAD. Whether circulating MPs contribute to impaired endothelial function and enhanced coagulation in patients with LVAD and thereby promote thrombotic complications is unknown.

The aims of this project are 1) to evaluate whether circulating MPs in patients with LVAD impair endothelial function and 2) to assess the procoagulative activity of circulating MPs in patients with LVAD in a prospective longitudinal study of patients undergoing LVAD implantation, 3) to analyze these parameters in the context of thromboembolic events.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: chronic heart failure INTERMASC 5-7 or
* Patients on LVAD support

Exclusion Criteria:

* current thrombembolic or bleeding event

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in the heart failure program of the University of Duesseldorf
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of thrombemboic events during 12 month | 12 month

SECONDARY OUTCOMES:
Endothelial function | Baseline
  Flow mediated dilatation measured by ultrasound
Level of circulating mircoparticles | Baseline
  measured and discriminated by FACS and ELISA
microparticle induced thrombin generation | Baseline
  measured and discriminated by FACS and ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Heinrich-Heine-University, Div. of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kramser N, Oehler D, Saeed D, Aubin H, Akhyari P, Kelm M, Westenfeld R, Horn P. Thromboembolic Events in Patients With Left Ventricular Assist Devices Are Related to Microparticle-Induced Coagulation. ASAIO J. 2021 Jan 1;67(1):59-66. doi: 10.1097/MAT.0000000000001200. PMID 33346991